CLINICAL TRIAL: NCT04154267
Title: Utility Evaluation of Protocolar Renal Transplant Biopsies in High Risk Patients for Immunological Loss of Graft
Brief Title: Protocol Biopsies in High-risk Renal Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20180625
Record Dates: First submitted 2019-10-21; First posted 2019-11-06 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant Failure; Kidney Transplant Infection; Kidney Transplant Failure and Rejection
Keywords: Kidney Transplantation; Protocol Biopsies; Kidney Transplant Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Intervention Model Description: We will include 100 patients in this work. In the first 48 hours after transplantation 50 patients will be randomized in the protocol biopsy and noninvasive evaluation group and 50 patients for noninvasive evaluation only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In addition to the routine evaluation commonly carried-out at this post-transplant period, protocol biopsies will be performed at the 10th-week post-transplantation in high-risk transplant recipients. Biopsy fragments will be evaluated for tissue immune aggression (mainly cellular and antibody-mediated rejections) and other conditions such as infections, particularly polyomavirus and cytomegalovirus and medication toxicities.
  Interventions: Procedure: Percutaneous renal biopsy.
- Control (No Intervention): Patients will only undergo routine noninvasive evaluation at this post-transplant period

INTERVENTIONS:
Procedure: Percutaneous renal biopsy. — The biopsy will be performed with a 16 Gauge semi-automatic needle gun for renal biopsy under real-time ultrasound control. After the procedure will be done ultrasound control
  Arms: Intervention

SUMMARY:
The present study aims to evaluate the usefulness of protocol biopsies in a cohort of renal transplant patients of high immunological risk for graft injury and loss.

DETAILED DESCRIPTION:
This will be a prospective study undertaken at the Renal Transplant Unit of Hospital of Clinics of Porto Alegre. In addition to the routine evaluation commonly carried-out at this post-transplant period, protocol biopsies will be performed at the 10th-week post-transplantation in high-risk transplant recipients. Biopsy fragments will be evaluated for tissue immune aggression (mainly cellular and antibody-mediated rejections) and other conditions such as infections, particularly polyomavirus and cytomegalovirus and medication toxicities. The presence of donor-specific antibodies and graft-damaging infectious agents will also be searched in the peripheral blood at the time of biopsy.One hundred patients will be randomized to a protocol biopsy and noninvasive assessment or only for noninvasive assessment. The hypothesis of the study is that biopsies will lead to treatments that may allow better outcomes of renal transplants, related to lowering the progression of subclinical aggressions, avoiding or delaying graft loss and preserving or decreasing the rate of loss of the glomerular filtration rate. Therefore, this strategy has the possibility of reaching clinical practice routine and thus contribute positively to the management of renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

Adult kidney transplants, with high immunological risk, who consented to participate in the study by signing the informed consent form. The high immune risk is defined by:

* Positive pre-transplant T-lymphocyte cross-test by flow cytometry (channel deviation greater than 62);
* Flow cytometry pre-transplantation positive B lymphocyte cross-test (channel deviation greater than 112);
* Calculated panel reactivity greater than 50% in class I and / or class II;
* Presence in the pre-transplantation serum of donor class I and / or II anti-Human Leukocyte Antigen antibodies with intensity and fluorescence greater than 1000;
* Occurrence of cellular or antibody-mediated rejection within 30 days prior to the date of the protocol biopsy.

Exclusion Criteria:

* Patients with contraindication to renal graft biopsy;
* Patients whose biopsy fragments are not representative;
* Patients with graft dysfunction in whom renal graft biopsy is indicated within 4 weeks prior to protocol biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of rejection. | Three months post transplant.
  To evaluate the incidence of subclinical, cellular and antibody-mediated rejections in protocol biopsies performed on patients at high immune risk who underwent kidney transplantation.

SECONDARY OUTCOMES:
Graft survival | Two years post transplant.
  Comparison of glomerular filtration rate at 2 years after transplantation between groups of patients with and without protocol biopsy using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Ceratti Manfro, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No